CLINICAL TRIAL: NCT00742456
Title: Insulin-induced Microvascular Dilatation During a Physiological Stimulus - Studies in Hypertension and Obesity.
Brief Title: Microvascular Dilatation After Endogenous Induced Hyperinsulinemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Prof. CDA Stehouwer, University Hospital Maastricht
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 08-2-031 MEC
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Hypertension; Obesity
Keywords: Microcirculation; Insulin; Hypertension; Obesity
MeSH Terms: conditions — Hypertension; Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Glucose
  Interventions: Dietary Supplement: Glucose solution
- II (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Glucose solution — single oral intake of 250 ml glucose solution (75gr sugar in 250ml of water)
  Arms: I
Dietary Supplement: Placebo — single intake of placebo solution (250ml of sweet flavored water, no sugar added), orally
  Arms: II

SUMMARY:
In this study we will examine if the insulin-induced microvascular effects will occur after a physiological stimulus (i.e. a oral glucose tolerance test). With that the physiological importance of the insulin-induced microvascular dilatation can be elucidated. In this study we hypothesize that oral glucose intake and consequently the endogenous induced hyperinsulinemia will lead to insulin-induced microvascular dilatation in healthy normotensive subjects. Furthermore, we suggest that the insulin-mediated microvascular dilatation, resulting from this physiological induced hyperinsulinemia, will be less in hypertensive and obese subjects compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

healthy normotensive subjects:

1. 18-60 years
2. Caucasian
3. Blood pressure <140/90 mmHg

obese normotensive subjects:

1. 18-60 years
2. Caucasian
3. Blood pressure <140/90 mmHg
4. BMI 30-38kg/m2

hypertensive subjects:

1. 18-60 years
2. Caucasian
3. Untreated hypertension >140/90mmHg.

Exclusion Criteria for healthy normotensive and hypertensive subjects:

1. Obesity (BMI>27kg/m2)
2. Cardiovascular disease (stroke, coronary artery disease, peripheral vascular disease, heart failure)
3. Diabetes mellitus according to the criteria of the ADA
4. Smoking
5. Alcohol use >4U/day
6. Use of medication (antihypertensive drugs, lipid lowering drugs, corticosteroids, NNSAIDs)
7. Pregnancy
8. Wearing contact lenses

for normotensive obese subjects:

1. Cardiovascular disease (stroke, coronary artery disease, peripheral vascular disease, heart failure)
2. Impaired glucose tolerance or diabetes mellitus according to the criteria of the ADA
3. Smoking
4. Alcohol use >4U/day
5. Use of medication (antihypertensive drugs, lipid lowering drugs, corticosteroids, NNSAIDs)
6. Pregnancy
7. Wearing contact lenses

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Functional recruitment of capillaries in the skin. | January 2009 - January 2010

SECONDARY OUTCOMES:
Perfused capillary density in the nailfold. | January 2009 - January 2010
Endothelium- (in)dependent vasodilatation of finger skin microcirculation | January 2009 - January 2010
Density of arterioles, capillaries and venules in the bulbar conjunctiva. | January 2009 - January 2010
Diameter of arterioles and venules in the bulbar conjunctiva. | January 2009 - January 2010
Insulin sensitivity (HOMA-IR) | January 2009 - January 2010

CONTACTS AND LOCATIONS:
Overall Officials: CDA Stehouwer, Prof., Study Chair — Univeristy Hospital Maastricht
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands